CLINICAL TRIAL: NCT03672708
Title: Cresyl Violet as a New Contrast Agent in Confocal Laser Endomicroscopy for in Vivo Diagnosis of Gastric Intestinal Metaplasia
Brief Title: Confocal Laser Endomicroscopy With Cresyl Violet for in Vivo Diagnosis of Gastric Intestinal Metaplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, vice president of Qilu Hospital, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018SDU-QILU-06
Record Dates: First submitted 2018-08-03; First posted 2018-09-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2018-09

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cresyl violet (Other)
  Interventions: Diagnostic Test: Cresyl violet

INTERVENTIONS:
Diagnostic Test: Cresyl violet — cresyl violet is applicated at the concentration of 0.15% via a spraying catheter to visualize cellular and tissue architecture in the pCLE

SUMMARY:
Confocal laser endomicroscopy (CLE) is a novel endoscopic system which can provide approximately 1000-fold magnification of the gastrointestinal mucosa. Previous studies have demonstrated its diagnostic value for Gastric intestinal metaplasia (GIM) with the use of a contrast agent.Recently, Cresyl violet (CV) has been used in CLE to visualize tissue architecture in human ileum, colon or myenteric plexus.No investigation has reported the characterization of GIM imaged with CLE when using CV as staining dye

ELIGIBILITY:
Inclusion Criteria:

* patients who had long-lasting upper gastrointestinal symptoms and aged 40 years or above
* patients with H. pylori infection, or known GIM or atrophic gastritis

Exclusion Criteria:

* patients with a history of GI surgery
* advanced gastric carcinoma or any other malignancy in the GI tract
* acute upper GI bleeding
* patients with contraindications to CLE examination, such as coagulopathy, pregnancy, breast feeding, impaired renal or liver function
* patients refused to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
feasibility of CV for identifying GIM | 1 month
  ratio of pCLE failure to visualize the cellular and subcellular structures
feasibility of CV for identifying GIM | 1 month
  ratio of pCLE failure to recognize lesions and their immediate characterization
newly pCLE criteria with CV application for GIM | 1 month
  ratio of diagnostic agreement between pCLE using CV and histopathological results
newly pCLE criteria with CV application for GIM | 1 month
  number of diagnostic agreement between pCLE with CV application and histopathological results

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD,MD, Study Director — Department of Gastroenterology,Qilu Hospital,shandong University; Zhen Li, PhD,MD, Study Director — Department of Gastroenterology,Qilu Hospital,shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China